CLINICAL TRIAL: NCT07268677
Title: A Single-arm Clinical Trial of Pirfenidone Plus Sintilimab Combined With Standard Neoadjuvant Chemotherapy for Patients With Colorectal Cancer Peritoneal Metastasis
Brief Title: A Single-arm Clinical Study Evaluating Pirfenidone and Sintilimab in Combination With Standard Neoadjuvant Chemotherapy for Colorectal Cancer Patients With Peritoneal Metastasis.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guoxiang Cai (Other)
Responsible Party: Sponsor-Investigator, Guoxiang Cai, Director, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDCRC0724
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pirfenidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pirfenidone plus sintilimab combined with standard neoadjuvant chemotherapy (Experimental)
  Interventions: Drug: pirfenidone plus sintilimab combined with standard neoadjuvant chemotherapy

INTERVENTIONS:
Drug: pirfenidone plus sintilimab combined with standard neoadjuvant chemotherapy — Treatment regimen: CapeOX + Pirfenidone + Sintilimab
  CapeOX:
  Oxaliplatin (L-OHP) 130 mg/m², IV infusion over 2 hours on Day 1 Capecitabine 1,000 mg/m² orally, twice daily for 14 consecutive days Repeated every 3 weeks
  Pirfenidone:
  Oral administration, 200 mg three times daily, taken on an empty stomach (low-dose regimen)
  Sintilimab:
  200 mg per dose, IV infusion once every 3 weeks The first 4 cycles are provided free of charge. After the fourth cycle, tumor response will be assessed; if continued use is required, a "buy 2, get 2 free" policy will apply.
  Tumor response evaluation will be performed after 4 treatment cycles.

SUMMARY:
Assuming that the objective response rate (ORR) of neoadjuvant chemotherapy in patients with colorectal cancer peritoneal metastasis is approximately 0.40 , a total sample size of 30 patients is required.

Step 1:

Ten patients will be initially enrolled. If the number of responders (CR/PR) is < 2, the study will be terminated early for futility.

If the number of responders is > 8, the treatment regimen will be considered effective, and the study may be concluded early.

Step 2:

If the number of responders in Step 1 is between 2 and 8, the study will continue to enroll an additional 20 patients until completion.

Treatment regimen: CapeOX + Pirfenidone + Sintilimab

CapeOX:

Oxaliplatin (L-OHP) 130 mg/m², IV infusion over 2 hours on Day 1 Capecitabine 1,000 mg/m² orally, twice daily for 14 consecutive days Repeated every 3 weeks

Pirfenidone:

Oral administration, 200 mg three times daily, taken on an empty stomach (low-dose regimen)

Sintilimab:

200 mg per dose, IV infusion once every 3 weeks The first 4 cycles are provided free of charge. After the fourth cycle, tumor response will be assessed; if continued use is required, a "buy 2, get 2 free" policy will apply.

Tumor response evaluation will be performed after 4 treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years;
2. Radiologically (CT/MRI/PET-CT/FAPI-PET) or pathologically confirmed peritoneal metastasis from colorectal cancer;
3. Planned to receive first-line chemotherapy;
4. ECOG performance status of 0-1;
5. Adequate hematologic, hepatic, and renal function:

   1. Neutrophil count ≥ 1.5 × 10⁹/L
   2. Platelet count ≥ 100 × 10⁹/L
   3. Hemoglobin ≥ 8.0 g/dL
   4. Creatinine clearance > 30 mL/min
   5. For patients without liver metastasis: AST and ALT ≤ 2.5 × upper limit of normal (ULN)
   6. Total bilirubin ≤ 2 × ULN
   7. APTT and PT ≤ 1.5 × ULN

Exclusion Criteria:

1. Individuals with a tendency to bleed, hereditary bleeding disorders, or evidence of coagulation abnormalities;
2. Pregnant or breastfeeding women, or women of childbearing potential who are not using effective contraception;
3. Expected survival ≤ 3 months;
4. Participation in another investigational drug trial within the past 4 weeks;
5. Prior treatment with any anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies (or any other antibodies targeting T-cell co-stimulation or immune checkpoint pathways);
6. Uncontrolled neurological or psychiatric disorders that may affect compliance or the ability to report treatment responses;
7. Known allergy to any study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 3months
  Objective Response Rate (ORR) is defined as the proportion of patients who achieve a best overall response of Complete Response (CR) or Partial Response (PR) during neoadjuvant therapy, as assessed by the investigator according to RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Overall survival | 2years
Safety | 6months
  The severity of adverse events was determined using the NCI-CTC AE 5.0 standard. During the trial, the adverse event record form should be filled in truthfully, including the time of occurrence, severity, relevance to the study treatment, duration, measures taken, and outcome of the adverse event.